CLINICAL TRIAL: NCT05672095
Title: Phase I/II Trial of Niraparib/Selenium Combination Treatment in Patients With BRCA1/2-Wild Type Recurrent Platinum-Resistant Ovarian Cancer
Brief Title: Niraparib and Selenium for the Treatment of Recurrent BRCA Negative Platinum Resistant Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Abandoned
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23231; NCI-2022-10203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20530 (Other: City of Hope Medical enter); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling; niraparib; Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selenium, niraparib) (Experimental): Patients receive selenium IV and niraparib PO on study. Patients also undergo CT, MRI, biopsy, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Niraparib; Other: Questionnaire Administration; Dietary Supplement: Selenium

INTERVENTIONS:
Procedure: Biopsy — Undergo needle or core biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827
Other: Questionnaire Administration — Ancillary studies
Dietary Supplement: Selenium — Given IV
  Other Names: Se

SUMMARY:
This phase I/II trial tests the safety, side effects and best dose of a combination therapy (niraparib and selenium) in treating patients with BRCA negative ovarian cancer that has come back (recurrent) and does not respond to platinum based therapy (platinum resistant). Selenium is a form of the trace element with potential antineoplastic activity which may help block the formation of growths that may become cancer. Niraparib is in a class of medications called poly (ADP-ribose) polymerase inhibitors. It works by killing cancer cells and helps maintain the response of certain types of ovarian, fallopian tube and peritoneal cancers. Giving selenium and niraparib may kill more cells in patients with ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety, tolerability and feasibility of administering niraparib/selenium combination therapy. (Phase I) II. To determine the anti-tumor activity of niraparib/selenium combination therapy, as assessed by median progression-free survival (PFS). (Phase II) III. To evaluate the tolerability of the combination therapy as assessed by a reduction in nausea, fatigue over historical rates. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the impact of treatment on quality of life over time, as evaluated by the Functional Assessment of Cancer Therapy - Ovarian Cancer (FACT-O) scores. (Phase I and Phase II) II. To estimate overall survival (OS), overall response rate (ORR), disease control rate (DCR), response duration and time to progression (TTP). (Phase I and Phase II)

CORRELATIVE OBJECTIVES:

I. To evaluate the molecular effects of selenium/niraparib combination therapy in ovarian tumors, as assessed by (Phase I and Phase II):

Ia. Changes in RAD51 foci formation which is a surrogate marker to examine homologous recombination by looking at tumor tissue prior to study and after 2 months of study therapy; Ib. By DNA full exome and RNA sequencing of tumors, protein profiling, prior to study and after 2 months of study therapy; Ic. Changes in RAD51AP1 expression in tumor tissue by Western blot prior to study and after 2 months of study therapy; Id. Changes in the endosomal vesicles (EV) markers in the urine, vaginal secretions, malignant effusions and plasma.

OUTLINE: This is a dose-escalation study of niraparib and selenium followed by a dose-expansion study. Patients are assigned to 1 of 2 phases.

Patients receive selenium intravenously (IV) and niraparib orally (PO) on study. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), biopsy, and collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from biopsy or tissue block cytology obtained at time of last disease recurrence. If biopsy is not possible or patient refuses, the principal investigator (PI) may allow an earlier biopsy to be tested. If unavailable, exceptions may be granted with Study PI approval
* Age: >= 18 years
* Eastern cooperative oncology group (ECOG) =< 2
* Histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal cancer. May not have non epithelial tumors or ovarian tumors with low malignant potential (ie, borderline tumors) or mucinous tumors or small cell carcinoma tumors or low grade serous carcinoma
* Recurrent, platinum resistant disease (defined as progression within <6 months from completion of platinum-based therapy. The date should be calculated from the last administered dose of platinum therapy)
* Measurable disease per response evaluation criteria in solid tumors (RECIST) 1.1 or evaluable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease related in the setting of CA125 >2x upper limit of normal [ULN])
* No more than 4 prior cytotoxic regimens (including primary therapy). Hormonal therapies (tamoxifen, aromatase inhibitors) or other prior poly (ADP-Ribose) polymerase (PARP) inhibitors will not count toward the prior regimen limit. Prior PARP inhibotor therapy is allowed
* Fully recovered from the acute toxic effects (except alopecia) to =< Grade 1 to prior anti-cancer therapy
* MyChoice HRD test should show BRCA wt and no HRD. No deleterious germline BRCA 1/2 mutations are allowed
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 150,000/mm^3 (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease, when =< 2.0 X ULN is acceptable (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN, unless liver metastases are present, in which case =< 5 x ULN (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN, unless liver metastases are present, in which case =< 5 x ULN (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Serum Creatinine =< 1.5 x ULN or creatine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Prothrombin (PT) =< 1.25 x ULN (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Hemoglobin >= 9 g/dL (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Women of childbearing potential (WOCBP): negative highly sensitive urine or serum pregnancy test (highly sensitive urine test will be required if serum pregnancy test is not available) (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Normal blood pressure or adequately controlled hypertension (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Agreement by subjects of childbearing potential* to use a highly effective method of birth control or abstain from heterosexual activity for the course of the study through at least 180 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, biological therapy, immunotherapy within 21 days prior to Day 1 of protocol
* Radiation therapy encompassing > 20% of the bone marrow within 2 weeks. Any radiation therapy within 1 week prior to Day 1 therapy
* Colony-stimulating factors (e.g. granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin within 4 weeks prior to day 1
* Receipt of a transfusion (platelets or red blood cells) within 4 weeks of D1
* Known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer in situ that has been definitively treated
* Strong CYP3A4 inducers/ inhibitors within 14 days prior to Day 1 of protocol therapy
* UGT1A1 inhibitors within 14 days prior to Day 1 of protocol therapy
* Herbal medications containing selenium within 14 days prior to Day 1 of protocol therapy
* Vitamin E within 14 days prior to Day 1 of protocol therapy
* Anticoagulants within 14 days prior to Day 1 of protocol therapy or active thromboembolism. The use of ASA or NSAIDS is allowed
* Live vaccines within 14 days prior to the first dose of study treatment. Seasonal flu vaccines that do not contain live viruses are allowed. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, bacille Calmette Guerin, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. Intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition (including aluminum) to study agent
* Hypersensitivity to any study agent, or its excipients, when administered alone
* History of Posterior Reversible Encephalopathy Syndrome (PRES)
* Issues with tolerating oral medication (e.g. inability to swallow pills, malabsorption issues, ongoing nausea or vomiting)
* Active diarrhea
* Clinically significant uncontrolled illness or medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric order that prohibits obtaining informed consent
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Major surgery (other than debulking or exploratory surgery for ovarian cancer) for any reason within 3 weeks prior to randomization and/or incomplete recovery from surgery
* Prior organ transplantation including allogenic stem cell transplantation
* Diagnosis of Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML)
* Known leptomeningeal disease, carcinomatous meningitis, or radiologic signs of CNS hemorrhage. Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable
* Active infections
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Patients must not have uncontrolled hypertension as defined by systolic blood pressure (SBP) >= 160mmHg or diastolic blood pressure (DBP) >= 90mmHg; patients whose blood pressure can be controlled medically are allowed to be rescreened once BP is under control
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-18 (Estimated); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (Phase I) | Up to 3 years
  Toxicity will be evaluated by adverse events. Observed toxicities will be summarized based on highest dose, severity, time of onset, duration, probable association with the study treatment and reversibility of outcome. For continuous variable, descriptive statistics (number [n], mean, standard deviation, standard error, median range will be provided.
Progression-free Survival (PFS) (Phase II) | From start of selenium treatment until date of death, relapse/progression, or last contact date, whichever comes first, assessed up to 3 years
  PFS will be estimated using the Kaplan-Meier product limit method.
Tolerability (Phase II) | Up to 3 years
  Tolerability will be assessed using the CTCAE 5.0. Reduction in percentage of patients experiencing nausea and fatigue.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  ORR to be evaluated by the proportion of patients with either a complete response or a partial response relative to the total number of patients.
Disease Control Rate | Up to 3 years
  Clinical benefit response is the best response recorded from start of treatment until disease progression/recurrence relative to the total number of patients.
Overall Survival (OS) | From start of treatment to date of death or last contact date, whichever comes first, assessed up to 3 years
  OS will be calculated using the Kaplan-Meier product limit method.
Response Duration | Up to 3 years
  Defined as the time from date of first documented response to documented disease relapse, progression or death whichever comes first.
Time to Progression | From the start of treatment to disease progression, assessed up to 3 years
Quality of Life (QOL) | Up to 3 years
  QOL will be measured using FACT-O questionnaire. Information will be tabulated and graphically displayed to describe the changes over time. For quantitative scales, data will be represented using means/medians, histogram and boxplots.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Rodriguez-Rodriguez, Principal Investigator — City of Hope Medical Center